CLINICAL TRIAL: NCT02705391
Title: A Pilot Study of the Utility of Perfusion MRI and MR Elastography for Surgical Planning, Radiotherapy Target Delineation, and Treatment Response Evaluation in Newly Diagnosed Ewing Sarcoma, Rhabdomyosarcoma and Soft Tissue Sarcoma Patients
Brief Title: Advanced MR Imaging in Sarcoma Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deanna H. Pafundi, Ph.D., Assistant Professor of Medical Physics, College of Medicine; Consultant Radiation Oncology Radiation Physics, Mayo Clinic
Other Study IDs: 15-005622
Record Dates: First submitted 2016-01-12; First posted 2016-03-10 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
We intend to investigate the clinical application of two emerging imaging modalities for which the technical capability is currently in place at Mayo Clinic. The treatment of Ewing Sarcoma (ES), Rhabdomyosarcoma (RMS) and soft tissue sarcoma (STS) patients on this study will involve multi-disciplinary contributions from nationally recognized sarcoma experts in Radiation Oncology, Radiology, Orthopedic Surgery, Pediatric Oncology, Medical Oncology and Pathology.

Patients will undergo additional magnetic resonance (MR) imaging at the same time as the standard imaging.

The ability to compare several imaging modalities within a single cohort of patients maximizes the potential of the study to impact the future management of sarcoma patients. The collaborative nature of this study, with essential contributions from many departments will undoubtedly improve the coordinated care of sarcoma patients and naturally disseminate the advanced imaging experience that is acquired.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 7 years.
* Histological confirmation of newly diagnosed localized or newly diagnosed with metastatic Ewing Sarcoma, Rhabdomyosarcoma or Soft tissue Sarcoma.
* Tumors > 5 cm in diameter.
* Planning to receive RT or surgery with or without adjuvant radiotherapy (RT) at Mayo Clinic Rochester.
* Provide informed written consent if ≥ 18 years. If < 18 years, provide informed written assent and parent or legal guardian provide informed written consent.
* Patients must have measurable disease as defined in Section 11.0.
* Willingness to participate in mandatory imaging studies at Mayo Clinic Rochester.
* Baseline MRE information deemed as acceptable for assessment
* Baseline perfusion MRI deemed as acceptable for assessment

Exclusion Criteria:

* Co-morbid conditions that would result in expected survival to be less than 5 years

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Histological confirmation of newly diagnosed localized or newly diagnosed with metastatic Ewing Sarcoma, Rhabdomyosarcoma or Soft tissue Sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Establish correlation between perfusion Magnetic Resonance imaging (MRI), 18F-flourodeoxyglucose (18F-FDG) PET activity, MRI contrast enhancement, Magnetic Resonance Elastography (MRE) | 5 years
Establish correlation between pathologic response for ES, RMS and STS | 5 years

SECONDARY OUTCOMES:
Establish a correlation between change in perfusion and tissue stiffness with event-free survival. | 5 years
Establish a correlation between change in perfusion and tissue stiffness with overall survival. | 5 years
Establish a correlation between change in perfusion and tissue stiffness with local control. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Pafundi, Ph D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials